CLINICAL TRIAL: NCT06273501
Title: Preoperative MRI and Magnetometer-guided Intraoperative Sentinel Lymph Node Detection With Superparamagnetic Iron Oxide Nanoparticles (SPIO) in Patients With Vulvar Cancer - a Feasibility Study (POSVUC Pilot)
Brief Title: MRI and Magnetometer-guided Sentinel Lymph Node Detection in Vulvar Cancer
Acronym: POSVUC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Katja Stenström Bohlin, Principal Investigator, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D-NR 2022-02876-01
Record Dates: First submitted 2024-02-07; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Vulvar Cancer; Lymph Node Metastasis
MeSH Terms: conditions — Vulvar Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Magtrace — Patients will receive superficial and interstitial injection with a 23 G needle with of a total volume of 0.1 - 1 ml Magtrace at four sites in or near the tumor in vulva, the same localization as the injections of Technetium99m and Patent blue for tracing SLNs performed at the surgery. The injection is performed by one of the gynecologic cancer surgeons participating in this study.The time of migration of SPIO to the groin nodes is not known for vulvar cancer. Transportation by dynamic MRI, with selective sequences repeated during a time span of 1- 60 minutes after the injection.

SUMMARY:
The aim of the feasibility study is to evaluate whether SPIO-MRI and a magnetometer could be a potential substitute to the routine dual technique in pre-and intraoperative SLN localization. Secondary, to explore if SPIO-MRI could predict lymph node status in comparison to histopathological analysis.

DETAILED DESCRIPTION:
Sentinel lymph node (SLN) biopsy is the routine procedure for nodal staging in early vulvar squamous cell carcinoma (VSCC) in the absence of clinical signs of lymph node metastasis. The gold standard technique for identifying SLN utilizes Technetium (Tc99m) lymphoscintigraphy and blue dye. An alternative method has emerged using superparamagnetic iron-oxide (SPIO) and magnetic resonance imaging (MRI).

This study aims to enroll 20 VSCC patients scheduled for the SLN procedure. Determination of the minimal dosage of SPIO required to avoid excessive MRI artifacts while still identifying the SLN. Intraoperative SLN detection with a magnetometer will be compared with the gold standard gamma probe.

As secondary objective, in addition to determining the SNL, MRI analysis of the nodal status will be evaluated for potential metastasis and compared to histopathological results.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed primary VSCC <4 cm, candidates for surgery with SLNB Age above 18

Signed and dated written consent before the start of specific protocol procedures.

ECOG performance status 0-2

Exclusion Criteria:

Contraindications for MRI such as electronic implants or severe claustrophobia

Hip replacement

Iron overload disease 4. Known hypersensitivity to iron or dextran compounds

Inability to understand given information and give informed consent or undergo study procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sentinel lymph node identification | Within 30 days after SPIO injection.
  The number of lymph nodes identified preoperatively with SPIO-enhanced MRI and intraoperatively with a magnetometer compared to Technetium-99m scintigraphy and blue dye.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Leonhardt, Principal Investigator — Department of radiology, Sahlgrenska University Hospital
Locations (1):
- Department of Obstetrics and gynecology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No